CLINICAL TRIAL: NCT05540314
Title: Robotic Bariatric Database (RBD) Collaborative
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 001.WMP.2022.D
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects that have undergone robotic bariatric surgery: Subjects that have undergone robotic bariatric surgery between January 2018 and December 2019
  Interventions: Procedure: robotic bariatric surgery

INTERVENTIONS:
Procedure: robotic bariatric surgery — robotic bariatric surgery

SUMMARY:
With increased prevalence of obesity in the general population over the past 30 years, researchers have been focused on the development of new treatment options to achieve long-lasting weight loss. In 1991, the National Institutes of Health Conference Statement on Gastrointestinal Surgery for Severe Obesity developed a consensus stating that bariatric surgery was the most effective treatment for obesity since it is associated with good long-term results in terms of weight loss, glycemic control and decreased mortality.

To collect and store clinical data related to the treatment outcomes of robotic bariatric surgery in order to develop an evidence base such that physicians can provide the best possible care to patients undergoing surgical weight loss interventions.

DETAILED DESCRIPTION:
With increased prevalence of obesity in the general population over the past 30 years, researchers have been focused on the development of new treatment options to achieve long-lasting weight loss.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Eligible for or have undergone robotic bariatric surgery per the treating physician
* Undergone robotic bariatric surgery between January 2018 and December 2019

Exclusion Criteria:

* Do not meet the Study Inclusion Criteria l

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 3. Undergone robotic bariatric surgery between January 2018 and December 2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Date of Birth | January 2018- December2019
  mm/dd/yyyy
Principal Operative Procedure is an Initial Primary Metabolic or Bariatric Procedure | January 2018- December 2019
  Yes or No
Patient has a history of metabolic or bariatric surgery | January 2018- December 2019
  Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Sachin S . Kukreja, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Charlton Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No